CLINICAL TRIAL: NCT01879930
Title: Chronic Bladder Pain Syndrome in Women: Can Doxycycline Help? A Prospective, Randomised,Placebo-controlled, Double-blind Study
Brief Title: Chronic Bladder Pain Syndrome in Women: Can Doxycycline Help? A Prospective Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 075/08; 2148 (Other: Inselspital); 2012DR4157 (Other: Swissmedic)
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Pelvic Pain Syndrome; Bladder Pain Syndrome
Keywords: randomized; placebo-controlled; double-blind study; doxycycline
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- doxycycline (Active Comparator): Zadorin-100® (doxycycline), licence number Swissmedic: 43051 Legal holder: Mepha Pharma AG, Aesch/BL
  Interventions: Drug: doxycycline
- placebo (Placebo Comparator): Placebo Galepharm Composition: lactose monohydrate, ceolus PH 102, croscarmellose sodium, magnesiumstearat, manufacturer: Pharmacy Hotz, 8700 Küsnacht, Switzerland
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: doxycycline — Zadorin-100® (doxycycline), licence number Swissmedic: 43051 Legal holder: Mepha Pharma AG, Aesch/BL
  Oral intake during study period (4 weeks) once in the morning and once in the evening
  The masking of the agents is conducted using bordeaux-coloured, opaque hard-gelatine capsules (size 00) of the French company LGA. The hard-gelatine capsules are each filled with 1 unit Zadorin® 100
  Other Names: Zadorin-100® (doxycycline), licence number Swissmedic: 43051
  Arms: doxycycline
Drug: placebo — Placebo Galepharm Composition: lactose monohydrate, ceolus PH 102, croscarmellose sodium, magnesiumstearat, manufacturer: Pharmacy Hotz, 8700 Küsnacht, Switzerland
  Oral intake during study period (4 weeks) once in the morning and once in the evening
  The masking of the agents is conducted using bordeaux-coloured, opaque hard-gelatine capsules (size 00) of the French company LGA. The hard-gelatine capsules are each filled with 1 unit placebo 100mg in the sham-group
  Other Names: Placebo Galepharm
  Arms: placebo

SUMMARY:
Chronic bladder pain syndrome is a chronic disabling disorder characterized by chronic pelvic pain, pressure or discomfort perceived to be related to the urinary bladder accompanied by at least one other urinary symptom such as persistent urgency or frequency in the absence of an identifiable cause. Chronic bladder pain syndrome severely decreases an individual's quality of life and represents a significant financial burden to those affected by it. Currently, multifactorial pathogenesis is assumed including endocrine-involvement, pelvic floor muscle irregularities, immunologic aspects and chemical causes. Corresponding to the wide spectrum of presumptive triggers, a large number of therapeutic approaches are propagated, however most are associated with limited effectiveness. Thus, treatment of BPS is a challenge and the ideal therapy remains to be elucidated. Microorganisms such as Chlamydia trachomatis, Ureaplasma urealyticum and Mycoplasma genitalium remains a challenge so that these organisms may well be involved in the pathogenesis of chronic bladder pain syndrome. The investigators hypothesise that doxycycline orally for 4 weeks, including therapy of the sexual partner, can significantly relieve symptoms in women with chronic bladder pain syndrome

DETAILED DESCRIPTION:
Background

Doxycycline is used to treat bacterial infections. Doxycycline is in a class of medications called tetracycline antibiotics. In addition to the general indications for all members of the tetracycline antibiotics group, doxycycline is frequently used to treat chronic prostatitis and pelvic inflammatory disease. Especially intracellular agents, such as chlamydia, are generally susceptible to doxycycline. Assuming this infection to be responsible for the chronic bladder pain syndrome in women, therapy will be performed in accordance with the authorised indication and dosage.Bacterial cystitis is an exclusion criterion for the diagnosis of chronic bladder pain syndrome. However, the detection of microorganisms such as Chlamydia trachomatis, Ureaplasma urealyticum and Mycoplasma genitalium remains a challenge so that these organisms may well be involved in the pathogenesis of chronic bladder pain syndrome. This is supported by the findings of our retrospective study1 that doxycycline orally for 4 weeks including therapy of the sexual partner lead to a reduction of symptoms in 71% of women complaining of persistent urgency and frequency, chronic urethral and/or bladder pain. Therefore, doxycycline therapy is sensible, especially considering that there are only a few, costly and often little effective symptomatic other treatment options.

Thus, we aim to investigate the effectiveness of doxycycline in women with chronic bladder pain syndrome in a prospective, randomised, placebo-controlled, double-blind study.

Chronic bladder pain syndrome is a chronic disabling disorder characterized by chronic pelvic pain, pressure or discomfort perceived to be related to the urinary bladder accompanied by at least one other urinary symptom such as persistent urgency or frequency in the absence of an identifiable cause2. In Europe, prevalence rates in women range from 306 to 450/100'0003,4 - much higher than previously estimated. Thus, chronic bladder pain syndrome is a serious economic problem for every health care system. In addition, chronic bladder pain syndrome severely decreases an individual's quality of life and represents a significant financial burden to those affected by it. Currently, multifactorial pathogenesis is assumed including endocrine-involvement, pelvic floor muscle irregularities, immunologic aspects and chemical causes. Corresponding to the wide spectrum of presumptive triggers, a large number of therapeutic approaches are propagated, however most are associated with limited effectiveness. Thus, treatment of BPS is a challenge and the ideal therapy remains to be elucidated. We hypothesise that doxycycline orally for 4 weeks, including therapy of the sexual partner, can significantly relieve symptoms in women with chronic bladder pain syndrome.

Objective

To proof or reject the effectiveness of doxycycline in treatment of chronic bladder pain syndrome

Methods

This is a prospective, randomised, placebo-controlled double-blind trial. Recruitment of the study participants is performed in the urologic outpatient clinic of University Hospital Inselspital Bern.

The randomisation-list in the institute of pharmacy University Hospital Inselspital Bern will only be accessible to unblinded employees. In case of unblinding an authorized member of the blinded trial team contacts the 24-hours service-number of the pharmacist on-duty in the institute of pharmacy. After disclosure of the patient-number, the pharmacist on-duty performs the unblinding and informs the authorized unblinded trial-member about allocation. Finally unblinding is registered on the randomization list by the pharmacist on-duty.

The unblinded trial-member will record the name of the person who performed unblinding and the date and reason for unblinding in the patient's medical record.

ELIGIBILITY:
Inclusion Criteria:

* Bladder pain / suprapubic pressure or discomfort for >6months
* Urgency/urgency incontinence and/or frequency for >6months
* Written informed consent (including confirmation that the partner will also be treated and that during the treatment period sexual intercourse is only allowed using condoms)

Exclusion Criteria

* age < 18 years
* Tetracycline allergy
* Intake of a tetracycline in the last 3 months
* pregnancy
* breast feeding
* bacterial cystitis in the last 4 weeks
* urethral/vaginal/cervical/uterine and/or rectal cancer
* chemical cystitis
* tuberculous cystitis
* benign or malignant bladder tumors
* Lack of radiologic exclusion of pelvic pathology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in the O'Leary-Sant IC symptom and problem index total score from baseline | 4, 8 , 24 weeks

SECONDARY OUTCOMES:
Changes of patient reported pain, urgency, frequency, functional bladder capacity documented in 72-hour pain and bladder diary, completed during the 3 days before the particular follow-up visit. | 4, 8, 24 weeks
Changes in sexual function assessed by the Female Sexual Function Index (FSFI) at the time of the particular follow-up visit | 4, 8, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Burkhard, Principal Investigator — Vice Chair urology dep. Inselspital; Claudia Meissner, MD, Study Chair — Department of Urology, Inselspital Bern
Locations (1):
- Dep. of Urology, Bern University Hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] van de Merwe JP, Nordling J, Bouchelouche P, Bouchelouche K, Cervigni M, Daha LK, Elneil S, Fall M, Hohlbrugger G, Irwin P, Mortensen S, van Ophoven A, Osborne JL, Peeker R, Richter B, Riedl C, Sairanen J, Tinzl M, Wyndaele JJ. Diagnostic criteria, classification, and nomenclature for painful bladder syndrome/interstitial cystitis: an ESSIC proposal. Eur Urol. 2008 Jan;53(1):60-7. doi: 10.1016/j.eururo.2007.09.019. Epub 2007 Sep 20. PMID 17900797
- [Result] Burkhard FC, Blick N, Hochreiter WW, Studer UE. Urinary urgency and frequency, and chronic urethral and/or pelvic pain in females. Can doxycycline help? J Urol. 2004 Jul;172(1):232-5. doi: 10.1097/01.ju.0000128698.93305.2e. PMID 15201781
- [Result] Temml C, Wehrberger C, Riedl C, Ponholzer A, Marszalek M, Madersbacher S. Prevalence and correlates for interstitial cystitis symptoms in women participating in a health screening project. Eur Urol. 2007 Mar;51(3):803-8; discussion 809. doi: 10.1016/j.eururo.2006.08.028. Epub 2006 Aug 30. PMID 16979286
- [Result] Leppilahti M, Tammela TL, Huhtala H, Auvinen A. Prevalence of symptoms related to interstitial cystitis in women: a population based study in Finland. J Urol. 2002 Jul;168(1):139-43. PMID 12050508
- [Result] O'Leary MP, Sant GR, Fowler FJ Jr, Whitmore KE, Spolarich-Kroll J. The interstitial cystitis symptom index and problem index. Urology. 1997 May;49(5A Suppl):58-63. doi: 10.1016/s0090-4295(99)80333-1. PMID 9146003